CLINICAL TRIAL: NCT02316093
Title: The Effects of Obesity on 8-Hydroxy-Deoxyguanosine Levels in Patients With and Without Periodontal Disease
Status: Completed | Type: Observational
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Figen ÖNGÖZ DEDE, Faculty of Dentistry, Bulent Ecevit University
Other Study IDs: 20136255051502
Record Dates: First submitted 2014-12-10; First posted 2014-12-12 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (6):
- obese-chronic periodontitis patients
  Interventions: Other: Procedure: Gingival Crevicular Fluid, Saliva and Blood Sampling
- obese-gingivitis patients
  Interventions: Other: Procedure: Gingival Crevicular Fluid, Saliva and Blood Sampling
- obese-periodontally healthy controls
  Interventions: Other: Procedure: Gingival Crevicular Fluid, Saliva and Blood Sampling
- normal weight-chronic periodontitis patients
  Interventions: Other: Procedure: Gingival Crevicular Fluid, Saliva and Blood Sampling
- normal weight-gingivitis patients
  Interventions: Other: Procedure: Gingival Crevicular Fluid, Saliva and Blood Sampling
- normal weight-periodontally healthy controls
  Interventions: Other: Procedure: Gingival Crevicular Fluid, Saliva and Blood Sampling

INTERVENTIONS:
Other: Procedure: Gingival Crevicular Fluid, Saliva and Blood Sampling

SUMMARY:
Obesity may affect periodontal health by inducing gingival oxidative damage through increased production in circulating reactive oxygen species (ROS). Several studies have demonstrated that 8-OHdG in bodily fluids can act as a biomarker of oxidative DNA damage in periodontal diseases and for evaluating the effect of periodontal treatment. In the present study we hypothesized that high ROS levels in circulation may increase oxidative stress levels in the gingival crevicular fluid (GCF) and saliva in obese patients with periodontal disease, thus periodontal therapy could have positive effects on ROS levels.

DETAILED DESCRIPTION:
The purpose of this study was to investigate the effects of obesity on 8-Hydroxy-deoxyguanosine (8-OHdG) levels in the bodily fluids of patients with and without periodontal disease and to evaluate changes after initial periodontal treatment.

Diagnosed as obese (n=45) and normal-weight (n=45) individuals were categorized; chronic periodontitis (CP), gingivitis (G) and periodontally healthy controls (CTRL). Gingival crevicular fluid (GCF), plasma, saliva samples and clinical measurements were obtained at baseline and a month after initial periodontal treatment.

Unstimulated salivary samples were collected using standard techniques. About 2 mL whole saliva was collected in disposable tubes and centrifuged immediately to remove cell debris (10,000 g x 10 minutes). The supernatants (50µL each) were stored at -40C until analyzed. GCF samples were collected from a mesio-buccal and disto-palatal site on each tooth (molars, premolars, canines/incisors). In the CP group, the samples were obtained from patients at areas with ≥5 mm CAL, ≥6 mm PD and ≥30% bone loss. In gingivitis group, GCF samples were obtained from teeth with BOP and without CAL. In the healthy group, GCF samples were collected from teeth exhibiting PD<3 mm without CAL and BOP. Six GCF samples were collected from each patient. The area was isolated with cotton rolls, saliva contamination elimination was ensured, and it was slightly air dried. GCF was sampled with paper strips. Paper strips were placed into the crevice until mild resistance was felt (intracrevicular method) and left in the position for 30 seconds. Strips contaminated with blood or saliva were discarded. Each sampled strip was placed into a 400µl eppendorf centrifuge tube and stored at -40C until analyzed.

Five milliliters of venous blood was taken from antecubital vein by using a standard venipuncture method. Obtained blood sample was collected in vacutainer tubes and anti-coagulated with EDTA. The blood samples were then stored at -40C until required for use in ELISAs.

Power analysis indicated that 12 individuals for each group would be sufficient to achieve 80% power to detect a difference of 0.05 between the alternative and the null hypotheses.

The Shapiro Wilk test was used to investigate whether or not the data were normally distributed. Continuous variables with unequal variances were compared by means of Welch and Tamhane's T2 post-hoc test for BMI, PD, CAL and the levels of 8-OHdG. The comparison of the age, GI, PI and BOP was analyzed using the Kruskal-Wallis non-parametric test followed by post hoc group comparisons with the Bonferroni-adjusted Mann-Whitney U test. Paired Student's t-test or Wilcoxon rank-sum test was used to compare the measurements at two points (baseline and after SRP). The Spearman's rank correlation test was also used to detect the relationship between biochemical and clinical findings.

ELIGIBILITY:
Inclusion Criteria:

* never-smokers
* no history of systemic disease
* no patients had been under periodontal treatment and medicine for at least 6 months before the study
* no pregnancy or lactation
* no alcohol or antioxidant vitamin consumption.

Exclusion Criteria:

-

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: a population who received periodontal treatment at the Periodontology Department
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
plasma, saliva and GCF levels of 8-OHdG | baseline
plasma, saliva and GCF levels of 8-OHdG | a month after periodontal treatment